CLINICAL TRIAL: NCT00099658
Title: Evaluation of Quantitative and Qualitative Antibody Responses to Streptococcus Pneumoniae and Haemophilus Influenzae Type b Conjugate Vaccines Amongst HIV-1-Exposed-Infected Children That Are Receiving Vs. Those Not Receiving Antiretroviral Therapy, as Well as Among HIV-1-Exposed-Uninfected Children and HIV-1-Unexposed-Uninfected Children
Brief Title: Safety of and Immune Response to a Pneumococcal Vaccine (PncCV) in HIV Infected and Uninfected Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CIPRA SA (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: James McIntyre, CIPRA-SA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIPRA-SA Project 4; U19AI053217 (NIH); CIPRA; Project 4
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections; Pneumococcal Infections
Keywords: MTCT
MeSH Terms: conditions — HIV Infections; Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): HIV-uninfected infants born to HIV-uninfected mothers
  Interventions: Biological: Pneumococcal polysaccharide-protein conjugate vaccine
- 2 (Experimental): HIV-infected infants in CDC Disease Category 1 who were randomly assigned to the delayed therapy arm (Arm 1) of CIPRA SA-Project 2
  Interventions: Biological: Pneumococcal polysaccharide-protein conjugate vaccine
- 3 (Experimental): HIV-infected infants in CDC Disease Category 1 who were randomly assigned to the first early therapy arm (Arm 2) of CIPRA SA-Project 2
  Interventions: Biological: Pneumococcal polysaccharide-protein conjugate vaccine
- 4 (Experimental): HIV-infected infants in CDC Disease Category 2 or 3 who were randomly assigned to the second early therapy arm (Arm 3) of CIPRA SA-Project 2
  Interventions: Biological: Pneumococcal polysaccharide-protein conjugate vaccine
- 5 (Experimental): HIV-uninfected infants born to HIV infected mothers
  Interventions: Biological: Pneumococcal polysaccharide-protein conjugate vaccine

INTERVENTIONS:
Biological: Pneumococcal polysaccharide-protein conjugate vaccine — Injection administered three times before the age of 24 weeks
  Other Names: PncCV

SUMMARY:
Infection by Streptococcal pneumoniae is a common invasive bacterial infection in HIV infected children. The purpose of this study is to determine the safety of and immune response to a pneumococcal polysaccharide-protein conjugate vaccine (PncCV) in HIV infected and uninfected children. The study will also determine the safety of and immune response to Haemophilus influenzae vaccine (HibCV) in these children. Recruitment for this study will occur at two hospitals in South Africa, and all HIV infected infants participating in this study must also be coenrolled in the CIPRA SA-Project 2 study.

DETAILED DESCRIPTION:
HIV infected children are at high risk for invasive pneumococcal disease (IPD) caused by the bacterium Streptococcus pneumoniae. Chemoprophylaxis has been used in children with certain diseases for the prevention of IPD, but drug resistance may develop with this prevention strategy. In contrast, a vaccine to prevent IPD would have fewer negative implications on future treatment options than chemoprophylaxis. This study will evaluate the safety of and immune response to PncCV in South African HIV infected and uninfected children. This study will also evaluate the safety of and immune response to HibCV in these children.

This study will last 5.5 years. There will be 5 groups in this study. Group 1 will be HIV uninfected infants born to HIV uninfected mothers. Group 2 will be HIV infected infants in CDC Disease Category 1 who were randomly assigned to the delayed therapy arm (Arm 1) of CIPRA SA-Project 2. Group 3 will be HIV infected infants in CDC Disease Category 1 who were randomly assigned to the first early therapy arm (Arm 2) of CIPRA SA-Project 2. Group 4 will be HIV infected infants in CDC Disease Category 2 or 3 who were randomly assigned to the second early therapy arm (Arm 3) of CIPRA SA-Project 2. Group 5 will be HIV uninfected infants born to HIV infected mothers; Group 5 infants will undergo repeat HIV testing at 4 to 8 months of age, 9 to 11 months of age, and approximately 18 months of age.

There will be 13 study visits; medical history assessment, a physical examination, and blood collection will occur at each visit. At each of 3 study visits before age 24 weeks, all participants will receive an injection of PncCV and an injection of routine pediatric vaccines, including HibCV. Previously vaccinated HIV infected participants will only receive those vaccines they need to complete the South African series of routine pediatric vaccinations. Within each group, participants will be randomly assigned to receive a booster shot of either PncCV or HibCV between 64 and 76 weeks of age. Participants will also receive two measles vaccinations between 38 and 76 weeks of age. Parents or guardians will be asked to complete a diary card after each vaccination and report any adverse effects occurring within the 72 hours post-vaccination.

ELIGIBILITY:
Inclusion Criteria for All Infants:

* Birth weight of at least 2 kg (4.4 lbs)
* Written informed consent from parent or guardian
* Mother's HIV status documented after 24th week of pregnancy, if her infant joins Group 5 and is HIV uninfected
* Parent or guardian of infant intends to remain in the study area for the duration of the trial

Inclusion Criteria for HIV Infected Infants:

* HIV infected
* Participating in CIPRA SA-Project 2

Exclusion Criteria for All Infants:

* Blood products prior to study entry
* Immunosuppressant agents for more than 2 weeks, within 1 week of study entry
* Unable to tolerate oral medications
* Presence of any major, life-threatening congenital defect
* Acute illness or fever requiring hospitalization within 72 hours of immunization
* Grade 2 vaccine-related allergic reaction
* Grade 3 or 4 clinical or laboratory toxicity related to vaccination
* Use of any antiretroviral therapies other than those allowed in CIPRA SA-Project 2. Infants who received antiretroviral drugs used to prevent mother-to-infant HIV transmission are eligible for this study.
* Use of investigational drugs, systemic cytotoxic chemotherapy, or interleukin or other immune modulators
* Require certain medications

Exclusion Criteria for HIV Uninfected Infants:

* Vaccines prior to study entry. Infants who have received bacille Calmette-Guerin or oral polio vaccines are not excluded.

Ages: 4 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 579 (Actual)
Dates: Start 2005-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Response rate to PncCV among children in Group 2 compared to those in Groups 1 and 3 | At Weeks 3 and 6
Response rate to PncCV among children in Group 2 compared to those in Groups 1 and 3 before receiving booster vaccine dose | At Weeks 64 through 76
Vaccine safety profiles after each of the three primary doses of PncCV and booster doses of PncCV and HibCV | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Shabir Madhi, MD, MBBCH, Mmed, FCPaeds, PhD, Study Chair — Chris Hani Baragwanath Hospital

REFERENCES:
- [Background] Klugman KP, Madhi SA, Huebner RE, Kohberger R, Mbelle N, Pierce N; Vaccine Trialists Group. A trial of a 9-valent pneumococcal conjugate vaccine in children with and those without HIV infection. N Engl J Med. 2003 Oct 2;349(14):1341-8. doi: 10.1056/NEJMoa035060. PMID 14523142
- [Background] Madhi SA, Kuwanda L, Cutland C, Holm A, Kayhty H, Klugman KP. Quantitative and qualitative antibody response to pneumococcal conjugate vaccine among African human immunodeficiency virus-infected and uninfected children. Pediatr Infect Dis J. 2005 May;24(5):410-6. doi: 10.1097/01.inf.0000160942.84169.14. PMID 15876939
- [Background] Madhi SA, Petersen K, Madhi A, Khoosal M, Klugman KP. Increased disease burden and antibiotic resistance of bacteria causing severe community-acquired lower respiratory tract infections in human immunodeficiency virus type 1-infected children. Clin Infect Dis. 2000 Jul;31(1):170-6. doi: 10.1086/313925. Epub 2000 Jul 25. PMID 10913417
- [Background] Nachman S, Kim S, King J, Abrams EJ, Margolis D, Petru A, Shearer W, Smith E, Moye J, Blanchard S, Hawkins E, Bouquin P, Vink P, Benson M, Estep S, Malinoski F; Pediatric AIDS Clinical Trials Group Study 292 Team. Safety and immunogenicity of a heptavalent pneumococcal conjugate vaccine in infants with human immunodeficiency virus type 1 infection. Pediatrics. 2003 Jul;112(1 Pt 1):66-73. doi: 10.1542/peds.112.1.66. PMID 12837869
- [Background] Pai VB, Heyneman CA, Erramouspe J. Conjugated heptavalent pneumococcal vaccine. Ann Pharmacother. 2002 Sep;36(9):1403-13. doi: 10.1345/aph.1A048. PMID 12196061
- [Derived] Mutsaerts EAML, Nunes MC, van Rijswijk MN, Klipstein-Grobusch K, Otwombe K, Cotton MF, Violari A, Madhi SA. Measles Immunity at 4.5 Years of Age Following Vaccination at 9 and 15-18 Months of Age Among Human Immunodeficiency Virus (HIV)-infected, HIV-exposed-uninfected, and HIV-unexposed Children. Clin Infect Dis. 2019 Aug 1;69(4):687-696. doi: 10.1093/cid/ciy964. PMID 30418528
- [Derived] Madhi SA, Izu A, Nunes MC, Violari A, Cotton MF, Jean-Philippe P, Klugman KP, von Gottberg A, van Niekerk N, Adrian PV; CIPRA 4 team. Longitudinal study on Streptococcus pneumoniae, Haemophilus influenzae and Staphylococcus aureus nasopharyngeal colonization in HIV-infected and -uninfected infants vaccinated with pneumococcal conjugate vaccine. Vaccine. 2015 May 28;33(23):2662-9. doi: 10.1016/j.vaccine.2015.04.024. Epub 2015 Apr 21. PMID 25910923
- See also: Click here for more information about CIPRA-SA Project 2. — http://clinicaltrials.gov/ct/show/NCT00102960